CLINICAL TRIAL: NCT02979808
Title: An Open, Qualitative, Prospective, Multicenter Trial of a Novel Transanal Irrigation System in Spinal Cord Injured Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply International (Industry)
Collaborators: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NAV-0001
Record Dates: First submitted 2016-11-07; First posted 2016-12-02 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Neurogenic Bowel
MeSH Terms: conditions — Neurogenic Bowel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Navina Smart (Experimental): Navina Smart will be used during 12 months for transanal irrigation (TAI).
  Interventions: Device: Navina Smart

INTERVENTIONS:
Device: Navina Smart — Subjects treatment-naïve to transanal irrigation (TAI). Frequency of TAI will be tailored to each subject.

SUMMARY:
This study is designed as an open, prospective, non-controlled, qualitative, multicentre study of a novel transanal irrigation system performed in a population of 150 subjects suffering from spinal cord injury and confirmed neurological bowel dysfunction. The study is expected to last for a total of 1 year (treatment period) with a planned 12- month recruitment period and three scheduled site visits.

DETAILED DESCRIPTION:
This study will be conducted in multiple countries, all outside of the United States. The study is approved by oversight authorities in the United Kingdom, Germany, Spain, Sweden, Denmark, Norway, France, and Italy

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent.
2. Male or female aged 18 years or older.
3. Patient with previously confirmed chronic spinal cord injury, either:

   1. Traumatic; at any level and any completeness of injury and ASIA grade classification, or
   2. Non-traumatic; due to infection, inflammation (i.e.; transverse myelitis or ischaemic myelitis), compromised blood supply, a post-ischemic state, etc.
4. At least 3 months post spinal cord injury at time of consent.
5. NBD score ≥10, confirmed at Baseline .
6. Only TAI treatment - naïve patient (not having previously used any particular transanal irrigation system, e.g. Peristeen®).
7. Confirmed NBD refractory to conservative therapy and judged eligible for transanal irrigation as per standardised treatment pathway 18.
8. Able to handle smartphone/tablet.

Exclusion Criteria:

1. Any confirmed or suspected diagnosis of anal or rectal stenosis, active inflammatory bowel disease, acute diverticulitis, severe diverticulosis, colorectal cancer, ischemic colitis, history of life-threatening autonomic dysreflexia, bleeding disorders, unspecified peri-anal conditions.
2. Untreated rectal impaction.
3. Any radiotherapy to the pelvis.
4. Any current treatment with anticoagulants (not including aspirin or clopidogrel).
5. Any current treatment with long-term systemic steroid medication (not including inhalation agents and/or local topical treatment).
6. Current use of prokinetics.
7. Any prior rectal or colonic surgery (not including anal procedures >3 months ago, e.g. haemorrhoid excision).
8. Anal, rectal and/or colonic endoscopic polypectomy within the previous 4 weeks.
9. Overt or planned pregnancy.
10. Ongoing symptomatic UTI as judged by investigator.
11. Diagnosed psychiatric illness, considered as unstable by the investigator.
12. Diagnosed with MS.
13. Involvement in the planning and conduct of the study (applies to both WHC staff and staff at the study site).
14. Previous enrolment in the present study.
15. Simultaneous participation in another clinical study that may interfere with the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in neurogenic bowel disfunction symptoms. | 3 months
  1. The primary objective of this study is to evaluate change in neurogenic bowel dysfunction symptoms between baseline and 3 months use of the Navina™ Smart system, as measured by a patient friendly version of the validated instrument NBD Score.

SECONDARY OUTCOMES:
Change of QoL status | Baseline, 3-months, 12-months
  To investigate the change of QoL status in the selected patient population (absolute values)
NBD symptoms | 6-months, 9-months, 12-months
  To investigate NBD symptoms after 6, 9 and 12 months use of Navina Smart system
Product use compliance. | 3-months, 6-months, 9-months, and 12-months
  Study product use compliance (is TAI still performed using the study device).
Patient satisfaction assessed through patient reported outcome (PRO) variables. | 3-months and 12-months
  To investigate patient perception and satisfaction of bowel management including TAI therapy and use of the Navina Smart system.
Frequency of urinary tract infection (UTI). | 3-months and 12-months
  Investigate frequency of UTI using patient reported outcome (PRO) variables.
Health economic analysis utilizing QoL data. | Baseline, 3-months, and 12-months.
  To perform health economic analyses using QoL data (EQ-5D).
Health economic analysis utilizing patient reported outcome (PRO) variables. | Baseline, 3-months, and 12-months.
  To perform health economic analyses using PRO variables.
Thematic analysis of interview data. | Baseline, 3-months, and 12-months (or at end of treatment period).
  To understand individual experience of initiating and using TAI for neurogenic bowel dysfunction.
Thematic analysis of interview data. | Baseline, 3-months, and 12-months (or at end of treatment period).
  To explore individual perceptions of using TAI compared with other conservative treatments for neurogenic bowel dysfunction.
Thematic analysis of interview data. | Baseline, 3-months, and 12-months (or at end of treatment period).
  To explore what influences individuals to continue with or stop using TAI for neurogenic bowel dysfunction.
Incidence of adverse events, serious adverse events, and adverse device effects. | 3-months, 6-months, 9-months, 12-months
  To evaluate short- and long-term safety of the product and therapy by assessing adverse events, serious adverse events, adverse device effects.

CONTACTS AND LOCATIONS:
Locations (11):
- Aarhus University Hospital, Aarhus, Denmark
- Hôpital St Jacques, Nantes, Rennes, France
- Germany (2):
  - Zentralklinik Bad Berka Gmbh, Bad Berka
  - BG-Klinikum Hamburg, Hamburg
- Italy (2):
  - Montecatone Rehabilitation Institute, Università di Bologna, Imola, Bologna
  - Azienda Ospedaliera- Universitaria Careggi, Florence, Florence
- Sunnaas Sykehus HF, Nesoddtangen, Norway
- Spain (2):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Unidad de Lesionados Medulares Hospital Traumatología, Barcelona
- Neurologiska kliniken, Avd R18 Karolinska Universitetssjukhuset, Solna, Stockholm, Sweden
- Gastrointestinal Physiology Unit, University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emmanuel A, Kurze I, Krogh K, Ferreiro Velasco ME, Christensen P, Del Popolo G, Bazzocchi G, Hultling C, Perrouin Verbe B, Bothig R, Glott T, Gonzalez Viejo MA. An open prospective study on the efficacy of Navina Smart, an electronic system for transanal irrigation, in neurogenic bowel dysfunction. PLoS One. 2021 Jan 29;16(1):e0245453. doi: 10.1371/journal.pone.0245453. eCollection 2021. PMID 33513187